CLINICAL TRIAL: NCT04415879
Title: Effects of a N95 Respirator vs Cloth Mask on Exercise Capacity During Treadmill Exercise.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Debasis Sahoo, Staff Physician, The Cleveland Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-538
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-05

CONDITIONS: COVID-19
Keywords: Exercise; Face Mask; COVID-19
MeSH Terms: conditions — COVID-19; Motor Activity | interventions — N95 Respirators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No Mask (Active Comparator): Individuals will perform a Modified Balke Treadmill test with no mask and their estimated VO2 peak will be calculated based off of peak workload.
  Interventions: Other: N-95 Respirator; Other: Cloth Face Mask
- N-95 Respirator (Experimental): Individuals will perform a Modified Balke Treadmill test while wearing a N-95 Respirator and their estimated VO2 peak will be calculated based off of peak workload.
  Interventions: Other: N-95 Respirator; Other: Cloth Face Mask
- Cloth Mask (Experimental): Individuals will perform a Modified Balke Treadmill test while wearing a cloth mask and their estimated VO2 peak will be calculated based off of peak workload.
  Interventions: Other: N-95 Respirator; Other: Cloth Face Mask

INTERVENTIONS:
Other: N-95 Respirator — N-95 mask will be worn as personal protective equipment during a graded exercise test
Other: Cloth Face Mask — A cloth mask will be worn as personal protective equipment during a graded exercise test

SUMMARY:
This study intends to find out how a cloth mask may impact exercise capacity, to provide guidance for exercisers to adjust their expectations and training accordingly. The investigators plan to asses exercise capacity through estimated peak oxygen consumption (eVO2peak), oxygen saturation and level of perceived exertion during treadmill based exercise while wearing a cloth mask compared to exercising without a cloth mask. The potential significance of this study is to determine if subjects can exercise safely and if their exercise training needs to be adjusted while following the current recommendations of wearing a cloth mask in public. The degree of airflow limitation experienced will depend on the type and fit of the mask being worn, and inadequeate airflow could possibly result in CO2 re-breathing if all air was not fully discharged from the mask with each breath. This re-breathing of CO2 could potentially limit the workload leading to a detriment in performance, and increase in adverse symptoms such as dizziness, lightheadedness, chest pain or shortness of breath that does not improve with rest.

DETAILED DESCRIPTION:
If healthcare providers are going to recommend that individuals exercise with cloth masks, it is imperative that future research is conducted to evaluate the degree to which airflow can be limited during exercise by wearing a cloth mask. At the completion of the study, the investigators will have further understanding of the effects of face masks during treadmill based running. To the investigators knowledge this is the first study to assess the effects of wearing protective cloth mask on exercise capacity.

Hypothesis The null hypothesis HO states that exercising with a cloth mask will be inferior to the current standard of exercising without a facemask, limiting peak exercise when non-inferiority margin is 1 estimated metabolic equivalent ( eMET 3.5 mlO2*kg-1*min-1).

The alternative hypothesis H1 states that exercising with a mask will not be inferior to the current standard of exercising without a facemask, limiting peak exercise when non-inferiority margin is 1 eMET.

EXPERIMENTAL DESIGN & METHODS Subject Recruitment: The investigators will recruit 20 subjects though the Cleveland Clinic. Inclusion Criteria: Healthy subjects age > 18, Exclusion Criteria: Any long-term disease that would interfere with their ability to exercise safely, fever >100.4 F, or pregnancy. Informed consent will be obtained by the CoPI, and need for medical clearance determined based on ACSM's 2015 preparticipation guidelines. To remain compliant with enterprise guidelines we will not be recruiting healthy subjects outside of the Cleveland Clinic staff at this time to avoid increase COVID-19 exposure risk. However, if the enterprise changes the guidelines we will expand our enrollment to include non Cleveland Clinic employees. Employees will not be solicited by direct initiation. Recruitment will involve only posted notice or general advertising that does not pressure employees into participating for fear of job loss, delayed promotion, or other influences from their superior.

Study Design: The study design is a prospective crossover non-inferiority trial where subjects will complete 3 separate graded exercise treadmill tests each time wearing either No Mask, N-95 Mask (3M), or Cloth Mask (Boco). The order of the mask worn will be randomly assign to minimize familiarization or training effect. All testing will be performed in a Cleveland Clinic facility following standardized COVID-19 screening precautions. The investigators will compare the data collected from each test to asses for differences between subject comfort, peak exercise capacity (eMET), heart rate response during exercise and recovery.

Testing: After completing the informed consent and being medically cleared, subjects will then perform a symptom limited graded exercise treadmill test using a modified Balke protocol with continuous 12-lead EKG monitoring. Exercise tests will be stopped if any significant cardiac arrhythmias occur or significant ST segment depressions develops. The test will be terminated if ST elevation (> 1.0 mm), marked ST displacement (horizontal or downsloping of > 2mm, measured 60 to 80 ms after the J point), moderate to severe angina, Signs of poor perfusion (cyanosis or pallor), Sustained ventricular tachycardia or other arrhythmia, including second or third decree AV block, that interferes with normal maintenance of cardiac output during exercise, or development of bunle-branch block that cnannot be distinguished from bentricular tachycardia. The modified Balke, which is a well-accepted treadmill protocol that keeps the speed constant and increases workload by grade. Subjects will rest for 3 minutes and resting heart rate, blood pressure, subjective perceptions of the face mask will be measured. Subjects then will walk at 0% grade at 3 miles per hour for 2 minutes. Elevation will be increased by 2% after the initial 2 minutes and by 1% each minute thereafter until the test is terminated. Heart rate, RPEand oxygen saturation will be measured with a pulse oximeter at baseline, last 5-10 seconds of each stage and the investigators will continue to monitor heart rate during recovery at 1, 3 and 5 minutes post exercise. The investigators will monitor each stage for perceived exertion, feelings of light headedness, anxiety, and discomfort. The test will also be terminated at the request of the subject or if any chest pain develops. The scale of measuring subjective perceptions instrument will be adminstereted after collecting 5 minutes of resting, end of the exercise test, and at 5 minutes post recovery. The graded exercise test will be performed once with No Mask, once with a 3M 8200 N-95 Respirator, and once with a Cloth Mask (Boco). Subjects will be randomized by a random number generater (1= No Mask, 2= N-95, 3= Cloth Mask) to determine the order the perform each exercise test No Mask, N-95 or Cloth Mask and will complete the other tests 2 atleast 1 day apart. Subjects will be instructed to abstain from exercise for 2 days before the test.

Mask:

3M 8200 N-95 Respirator obtain from a third party provider. N-95 Respirators have been purchased outside the Cleveland Clinic supply chain. Cloth Face Mask manufactured by Boco is a custom designed two-layer face masks are built with a tightly woven polyester outer shell fabric and a soft, breathable performance knit mesh inner linig. Includes a slit pocket where a filter can be added.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Cleveland Clinic Employee
* Must not be pregnant

Exclusion Criteria:

* Medical condition that would interfere with ability to exercise safely

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | 4 Weeks
  To gain further understanding on effects exercising with a cloth mask has on exercise capacity. Our working hypothesis is that wearing a face mask will limit exercise capacity by a minimal clinically important difference (MCID) of 1 estimated Metabolic Equivalent (eMET 3.5 O2 ml/kg/min).

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No